CLINICAL TRIAL: NCT06512077
Title: Clinical Validation of Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Non-invasive Blood Glucose Detection in Non-diabetic Subjects
Brief Title: Clinical Validation of mμSORS for Non-invasive Blood Glucose Detection in Non-diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Photonic View Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCEMD20240701
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Validation of mμSORS for Noninvasive Blood Glucose Detection in healthy subjects (Experimental): Enrolled subjects will perform oral glucose tolerance test or hyperinsulin-hypoglucose clamp test. A measurement session of blood glucose consists of plasma sample and a measurement by mμSORS will be conducted synchronously.
  Interventions: Device: Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection

INTERVENTIONS:
Device: Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection — Blood glucose of participants were measured by venous plasma and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS). The two measurements were collected synchronously and analyzed.

SUMMARY:
This is a single-center, open-label, prospective study. Blood glucose is measured at different time points during oral glucose tolerance test and hypoglucose clamp test in healthy subjects, using both venous plasma and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS). Venous plasma glucose was set as gold standard. The two measurements were collected synchronously so as to calculate the mean absolute relative difference (MARD) and the consensus error grid (CEG). Accuracy of non-invasive blood glucose testing by mμSORS will be in-depth validated specifically in the 3-10 mmol/l glucose range.

DETAILED DESCRIPTION:
In order to clinically verify the accuracy and safety of non-invasive blood glucose measurement by the mμSORS technology specifically in the 3-10 mmol/l glucose range, this study will conduct oral glucose tolerance tests and hypoglucose clamp tests on healthy subjects at different time points during the tests. In oral glucose tolerance tests, there will be 9 points as follows: 0-min and post glucose-load 30-min, 60-min, 90-min, 120-min, 150-min, 180-min, 210-min and 240-min. While in hypoglucose clamp tests, blood glucose will be set at around 3.0-4.0mmol/l for about 1.5-2.0 hours, blood glucose will be detected every 10 minutes.

ELIGIBILITY:
Inclusion Criteria :

* Male or female.
* Aged>=18 years for OGTT participants or aged between 20 and 40 years for hypoglucose clamp tests participants.
* Fasting blood glucose (FPG) < 6.1 mmol/L and glycated hemoglobin (HbA1c) < 5.7% during the screening period.
* There are no scars, obvious pigmentation and other factors that interfere with the detection of the palm skin to be tested.
* Confirmed as healthy based on the results of physical examination, medical history, vital signs and clinical laboratory tests.
* Fully understand the nature, significance, possible benefits, possible inconveniences or potential risks of this research, and should also understand the research procedures, be willing to complete the entire research process, and provide written consent form.

Exclusion Criteria :

* With diabetes history.
* Any history of serious clinical diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry or metabolic abnormality, or any other disease that can interfere with the test results, which the investigator considers significant.
* Alcohol dependency or drug abuse.
* Those who have participated in clinical trials of other drugs within 3 months before screening (since the last visit of the previous trial).
* Those who have used any drugs that affect blood glucose levels (such as insulin, oral hypoglycemic drugs, steroid hormones, thyroxine, etc.) within 28 days before screening;
* Pregnancy or lactation period.
* Difficulty in venous blood collection or fainting of needles or blood.
* Other circumstances that the investigator considers inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative deviation (MARD) of venous plasma glucose and glucose values measured by mμSORS at each time point of OGTT and hypoglucose clamp tests. | 2 months
  Glucose will be measured using both intravenous sampling (plasma) and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS) detection synchronously.
Consensus Error Grid (CEG) for venous plasma glucose and glucose values measured by mμSORS at each time point of OGTT and hypoglucose clamp tests. | 2 months
  Glucose will be measured using both intravenous sampling (plasma) and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS) detection synchronously.

SECONDARY OUTCOMES:
MARD for two measurement methods in different blood glucose ranges. | 2 months
  Plasma glucose ranges 3.9-10.0 mmol/L and <3.9 mmol/L.
Incidence of Treatment-Emergent Adverse Events. | 2 months
  Safety outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China